CLINICAL TRIAL: NCT01931475
Title: Effect of Duloxetine 60mg Once Daily in Patients With Chronic Pain Due to Osteoarthritis in China
Brief Title: A Study of Duloxetine in Participants With Chronic Pain Due to Osteoarthritis in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13494; F1J-MC-HMGS (Other: Eil Lilly and Company)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): Double Blind Treatment Phase:
  60 milligram (mg) duloxetine administered by mouth once a day (QD). Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD for 12 weeks.
  Extension Treatment Phase:
  60 mg duloxetine administered by mouth QD for 13 weeks.
  Taper Phase: 1-week taper where participants taking 60 mg QD duloxetine during the study had their dosage reduced to 30 mg to minimize discontinuation-emergent adverse events (DEAEs).
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Double Blind Treatment Phase:
  Placebo administered by mouth once a day (QD) for 13 weeks.
  Extension Treatment Phase:
  60 mg duloxetine administered by mouth QD for 13 weeks. Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD.
  Taper Phase: 1-week taper - Placebo administered for 1 week if the participant discontinued from double blind treatment phase, or duloxetine 30 mg QD administered for 1 week if the participant discontinued from extension treatment phase or completed treatment. 1 week taper is to minimize discontinuation-emergent adverse events (DEAEs).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of duloxetine once daily compared with placebo on the reduction of pain due to osteoarthritis (OA) in knee or hip in participants in China.

ELIGIBILITY:
Inclusion Criteria:

* Meet clinical and radiographic criteria for the diagnosis of OA of the knee or hip with pain for ≥14 days of each month for 3 months prior to study entry
* Have a rating ≥4 on the Brief Pain Inventory (BPI) 24-hour average pain item (Question 3 of the BPI modified short form) at both Screening and Randomization

Exclusion Criteria:

* Have previously completed/withdrawn from this study or any other study investigating duloxetine (Note: Participants who have been previously screened for a duloxetine study other than this study and never received investigational product will be eligible for this study if they meet all current entry criteria)
* Have had previous exposure to duloxetine
* Have any previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder
* Current (within 1 year of Screening) Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Axis I diagnosis of major depressive disorder, anxiety disorders (excluding phobias), alcohol or eating disorders, as determined by the Mini-International Neuropsychiatric Interview or a previous diagnosis
* Have a history of substance abuse or dependence within the past year, excluding nicotine and caffeine
* Are taking any excluded medications that cannot be discontinued at Screening
* Have had treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization or the potential need to use an MAOI during the study or within 5 days of discontinuation of investigational product
* Have a positive urine drug screen for any substance of abuse or excluded medication
* Have serious cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study
* Have a history of recurrent seizures other than febrile seizures
* Are judged clinically by the investigator to be at suicidal risk according to the Columbia - Suicide Severity Rating Scale (C-SSRS): a "Yes" answer to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the"Suicidal Ideation" portion of the C-SSRS or a "Yes" answer to any of the suicide related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "Suicidal Behavior" portion of the C-SSRS, with the ideation/behavior having occurred within the previous month
* Have uncontrolled narrow-angle glaucoma
* Have acute liver injury (such as hepatitis) or severe cirrhosis
* Have known hypersensitivity to duloxetine or any of the inactive ingredients or have frequent/severe allergic reactions to multiple medications
* Have frequent falls that could result in hospitalization or could compromise response to treatment
* Have a diagnosis of inflammatory arthritis [that is, rheumatoid arthritis (RA)] or an autoimmune disorder (excluding inactive Hashimoto's thyroiditis)
* Have received intra-articular hyaluronate/steroids, joint lavage, or other invasive therapies to the index joint in the previous 3 months
* Have had arthroscopy of the index joint within the previous year or joint replacement of the index joint at any time
* Have surgery of the index joint scheduled to occur during the trial or are anticipated by the investigator to require surgery for the treatment of the OA of the index hip or knee along the duration of the study
* Have had a prior synovial fluid analysis showing a white blood cell (WBC) count ≥2000 cubic millimeter (mm3) that is indicative of a diagnosis other than OA
* Are non-ambulatory or require the use of crutches or a walker
* Have a body mass index >40
* Are anticipated by the investigator to require use of analgesic agents including, but not limited to, nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen/paracetamol, and opioids, or other excluded medication for the duration of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eil Lilly and Company
Locations (12):
- China (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bengbu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pingxiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tianjin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhuzhou

REFERENCES:
- [Derived] Leaney AA, Lyttle JR, Segan J, Urquhart DM, Cicuttini FM, Chou L, Wluka AE. Antidepressants for hip and knee osteoarthritis. Cochrane Database Syst Rev. 2022 Oct 21;10(10):CD012157. doi: 10.1002/14651858.CD012157.pub2. PMID 36269595
- [Derived] Yue L, Wang J, Enomoto H, Fujikoshi S, Alev L, Cheng YY, Skljarevski V. The Clinical Relevance of Pain Severity Changes: Is There Any Difference Between Asian and Caucasian Patients With Osteoarthritis Pain? Pain Pract. 2020 Feb;20(2):129-137. doi: 10.1111/papr.12835. Epub 2019 Nov 20. PMID 31505082
- [Derived] Wang G, Bi L, Li X, Li Z, Zhao D, Chen J, He D, Wang CN, Wu T, Duenas H, Skljarevski V, Yue L. Maintenance of effect of duloxetine in Chinese patients with pain due to osteoarthritis: 13-week open-label extension data. BMC Musculoskelet Disord. 2019 Apr 22;20(1):174. doi: 10.1186/s12891-019-2527-y. PMID 31010413
- [Derived] Yue L, Luo S, Wang Y, Wang CN, Duenas HJ, Skljarevski V. Clinical meaningfulness of duloxetine's effect in Chinese patients with chronic pain due to osteoarthritis: post hoc analyses of a phase 3 randomized trial. Open Access Rheumatol. 2019 Mar 21;11:67-76. doi: 10.2147/OARRR.S193044. eCollection 2019. PMID 30962729
- [Derived] Wang G, Bi L, Li X, Li Z, Zhao D, Chen J, He D, Wang CN, Duenas H, Skljarevski V, Yue L. Efficacy and safety of duloxetine in Chinese patients with chronic pain due to osteoarthritis: a randomized, double-blind, placebo-controlled study. Osteoarthritis Cartilage. 2017 Jun;25(6):832-838. doi: 10.1016/j.joca.2016.12.025. Epub 2016 Dec 31. PMID 28043937

RESULTS

PARTICIPANT FLOW:
Groups:
- 60 mg Duloxetine: Double Blind Treatment Phase:
  60 milligram (mg) duloxetine administered by mouth once a day (QD). Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD for 12 weeks.
  Extension Treatment Phase:
  60 mg duloxetine administered by mouth QD for 13 weeks.
  Taper Phase: 1-week taper where participants taking 60 mg QD duloxetine during the study had their dosage reduced to 30 mg to minimize discontinuation-emergent adverse events (DEAEs).
- Placebo: Double Blind Treatment Phase:
  Placebo administered by mouth once a day (QD) for 13 weeks.
  Extension Treatment Phase:
  60 mg duloxetine administered by mouth QD for 13 weeks. Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD.
  Taper Phase: 1-week taper - Placebo administered for 1 week if the participant discontinued from double blind treatment phase, or duloxetine 30 mg QD administered for 1 week if the participant discontinued from extension treatment phase or completed treatment.1 week taper is to minimize discontinuation-emergent adverse events (DEAEs).
Period: Period 1: Double-Blind Treatment Phase
Arm/Group | 60 mg Duloxetine | Placebo
Started | 205 | 202
Received at Least 1 Dose of Study Drug | 199 | 198
Completed | 166 | 176
Not Completed | 39 | 26
Not completed — Adverse Event | 20 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 16 | 12
Not completed — Lack of Efficacy | 2 | 3
Not completed — Physician Decision | 0 | 1
Period: Period 2: Extension Treatment Phase
Arm/Group | 60 mg Duloxetine | Placebo
Started | 166 | 176
Received at Least 1 Dose of Study Drug | 166 | 175
Completed | 162 | 157
Not Completed | 4 | 19
Not completed — Adverse Event | 0 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Study Terminated by Sponsor | 1 | 0
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 mg Duloxetine | Placebo | Total
Number analyzed (Participants) | 205 | 202 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.17 (8.19) | 59.83 (8.40) | 61.14 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 151 | 311
  Male | 45 | 51 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 205 | 202 | 407
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 205 | 202 | 407

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Brief Pain Inventory (BPI) 24-hour Average Pain Score
Description: BPI is a self-reported scale that measures the severity of pain based on the average pain during the past 24-hours. The severity scores ranged from 0 (no pain) to 10 (pain as severe as you can imagine). Least squares (LS) mean was calculated using mixed model repeating measures (MMRM) and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 172 | 177
units on a scale | -2.23 (0.11) | -1.73 (0.11)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.80 to -0.2]

2. Secondary Outcome: Patient Global Impressions of Improvement (PGI-I) Score
Description: PGI-I measures a participant's perception of improvement at the time of assessment compared with the start of treatment. Score ranges from 1 (very much better) to 7 (very much worse). Least squares (LS) mean was calculated using mixed model repeating measures (MMRM) and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: 13 Weeks
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 172 | 177
units on a scale | 2.73 (0.07) | 3.09 (0.07)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.54 to -0.19]

3. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Total and Subscale Scores
Description: WOMAC consists of 24 items divided into 3 subscales:Pain(5 items):during walking,using stairs,in bed,sitting or lying,and standing Stiffness;(2 items):after first waking and later in the day Physical Function;(17 items):stair use,rising from sitting, standing, bending,walking,getting in/out of a car,shopping,putting on/taking off socks,rising from bed,lying in bed,getting in/out of bath,sitting,getting on/off toilet,heavy household duties,light household duties.Each question is answered using a 5-point Likert scale(0 to 4).Pain subscale has a range of scores of 0(none) to 20(extreme).Stiffness subscale has a range of scores of 0(none) to 8(extreme).Physical function subscale has a range of scores of 0(none) to 68(extreme).Total score ranges from 0(none) to 96(extreme).Least squares(LS) mean was calculated using analysis of covariance(ANCOVA) and adjusted for treatment, pooled investigator,and baseline score.Last observation carried forward (LOCF) method was be used for these analyses.
Time Frame: Baseline, Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 184 | 182
units on a scale
  Total Score | -13.58 (0.92) | -10.09 (0.90)
  Pain | -3.03 (0.21) | -2.32 (0.21)
  Physical Function | -9.64 (0.68) | -7.28 (0.67)
  Stiffness | -0.83 (0.10) | -0.44 (0.10)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -3.49, 95% CI 2-sided [-5.62 to -1.35] — Total Score
Statistical Analysis 2: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.21 to -0.21] — Pain
Statistical Analysis 3: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -2.36, 95% CI 2-sided [-3.95 to -0.78] — Physical Function
Statistical Analysis 4: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.62 to -0.16] — Stiffness

4. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score
Description: CGI-S measures severity of illness at the time of assessment compared with start of treatment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least squares (LS) mean was calculated using mixed model repeating measures (MMRM) and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: Baseline,13 Weeks
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 172 | 177
units on a scale | -0.81 (0.05) | -0.53 (0.05)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.41 to -0.15]

5. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Severity
Description: BPI Severity of Worst Pain is self-reported scale that measures the severity of pain based on the worst pain experienced during the past 24-hours. The severity scores ranged from 0 (no pain) to 10 (pain as severe as you can imagine). BPI Severity of Least Pain is a self-reported scale that measures the severity of pain based on the least pain experienced during the past 24-hours. The severity scores ranged from 0 (no pain) to 10 (pain as severe as you can imagine). BPI Severity of Right Now Pain is a self-reported scale that measures the severity of pain based on the pain right now. The severity scores ranged from 0 (no pain) to 10 (pain as severe as you can imagine). Least squares (LS) mean was calculated using mixed model repeating measures (MMRM) and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 172 | 177
units on a scale
  BPI Severity of Worst Pain | -2.71 (0.14) | -2.00 (0.14)
  BPI Severity of Least Pain | -1.48 (0.12) | -1.20 (0.12)
  BPI Severity of Right Now Pain | -2.21 (0.14) | -1.74 (0.13)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.07 to -0.34] — BPI Severity of Worst Pain
Statistical Analysis 2: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.60 to 0.03] — BPI Severity of Least Pain
Statistical Analysis 3: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.82 to -0.11] — BPI Severity of Right Now Pain

6. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Interference
Description: BPI Interference Average Score is a self-reported scale that measures interference of pain on average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people,sleep, and enjoyment of life.The average Interference scores ranged from 0 to 10. General activity, mood,walking ability, normal work,relations with other people, sleep and enjoyment of life is each is a self-reported scale that measures the interference of pain in the past 24 hours on general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life.The Interference scores ranged from 0 (does not interfere) to 10 (completely interferes).Least squares (LS) mean was calculated using mixed model repeating measures (MMRM) and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 172 | 177
units on a scale
  BPI Interference Average Score | -1.63 (0.10) | -1.36 (0.10)
  General activity | -2.39 (0.14) | -1.83 (0.14)
  Mood | -1.43 (0.13) | -1.04 (0.13)
  Walking ability | -2.35 (0.14) | -1.88 (0.13)
  Normal work | -2.06 (0.14) | -1.76 (0.14)
  Relations with other people | -0.90 (0.11) | -0.84 (0.11)
  Sleep | -1.21 (0.14) | -0.99 (0.13)
  Enjoyment of life | -1.14 (0.13) | -1.07 (0.13)
Statistical Analysis 1: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.53 to -0.02] — BPI Interference Average Score
Statistical Analysis 2: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.94 to -0.19] — General activity
Statistical Analysis 3: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.74 to -0.05] — Mood
Statistical Analysis 4: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Median Difference (Final Values) = -0.47, 95% CI 2-sided [-0.82 to -0.11] — Walking ability
Statistical Analysis 5: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Median Difference (Final Values) = -0.31, 95% CI 2-sided [-0.68 to 0.06] — Normal work (includes both work outside the home and housework)
Statistical Analysis 6: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.34 to 0.21] — Relations with other people
Statistical Analysis 7: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.57 to 0.14] — Sleep
Statistical Analysis 8: Comparison: 60 mg Duloxetine vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.40 to 0.27] — Enjoyment of life

7. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale-Depression (HADS-D) or HADS-Anxiety (HADS-A) Subscale Scores
Description: HADS is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item was rated on a 4-point scale [0 (low level of anxiety or depression) to 3 (high level of anxiety or depression)], giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale were considered to be a 'significant' case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.' Mean was calculated using analysis of covariance (ANCOVA) and adjusted for treatment, pooled investigator, and baseline score. The last observation carried forward (LOCF) method will be used for these analyses.
Time Frame: Baseline, Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 182 | 182
units on a scale
  Depression Subscale | -0.10 (2.05) | -0.10 (2.12)
  Anxiety Subscale | 0.02 (2.58) | 0.08 (2.42)

8. Secondary Outcome: Change in Brief Pain Inventory (BPI) Average Pain Intensity Scores, Hospital Anxiety and Depression Scale (HADS) Depression Subscale (HADS-D) and HADS Anxiety Subscale (HADS-A)
Description: Evaluation on whether the change in BPI average pain intensity scores is a direct analgesic effect of duloxetine and is independent of treatment effect on mood, as measured by Hospital Anxiety and Depression Scale (HADS) depression subscale (HADS-D), or anxiety as measured by HADS anxiety subscale (HADS-A). Path analysis for the direct analgesic effect was used to test the null hypothesis that the change in BPI average pain severity depends on the improvement of HADS-D or HADS-A, versus the alternative that the improvement in BPI average pain severity is due to a direct analgesic effect of the treatment and not dependent upon the improvement in depression and anxiety symptoms.
Time Frame: Baseline, Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Participants (60 mg Duloxetine & Placebo): Duloxetine:
  Double Blind Treatment Phase:
  60 milligram (mg) duloxetine administered by mouth once a day (QD). Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD for 12 weeks.
  Extension Treatment Phase:
  60 mg duloxetine administered by mouth QD for 13 weeks.
  Taper Phase: 1-week taper where participants taking 60 mg QD duloxetine during the study had their dosage reduced to 30 mg.
  Placebo:
  Double Blind Treatment Phase:
  Placebo administered by mouth once a day (QD) for 13 weeks.
  Extension Treatment Phase:
  60 mg duloxetine administered by mouth QD for 13 weeks. Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD.
  Taper Phase:
  1-week taper - Placebo administered for 1 week if the participant discontinued from double blind treatment phase, or duloxetine 30 mg QD administered for 1 week if the participant discontinued from extension treatment phase or completed treatment.
Arm/Group | All Participants (60 mg Duloxetine & Placebo)
Number analyzed (Participants) | 364
units on a scale
  BPI average pain score | -1.91 (1.52)
  HADS-Depression subscale score | -0.10 (2.08)
  HADS-Anxiety subscale score | 0.05 (2.50)
Statistical Analysis 1: Comparison: All Participants (60 mg Duloxetine & Placebo); Path analysis for the direct analgesic effect was used to test the null hypothesis that the change in BPI average pain severity depends on the improvement of HADS-D or HADS-A, versus the alternative that the improvement in BPI average pain severity is due to a direct analgesic effect of the treatment and not dependent upon the improvement in depression and anxiety symptoms; Test type: Superiority or Other; p = 0.002, Regression, Linear; Total Effect = 97.49

9. Secondary Outcome: Percentage of Participants With Reduction of ≥30% and ≥50% in BPI Average Pain Score
Description: Pain severity was measured using an 11 point BPI scale from 0 (no pain) to 10 (worst pain) to determine average pain in the past 24 hours (average pain). A 30% (or 50%) improvement was defined as a ≥30% (or ≥50%) reduction in BPI pain severity from baseline to endpoint. Percentage of participants = (number of participants with ≥30% or ≥50% pain reduction / total number of participants in treatment group) * 100.The last observation carried forward (LOCF) method will be used for these analyses.
Time Frame: Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Number; unit: percentage of participants
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 194 | 197
percentage of participants
  Participants with >=30% Reductions | 63.40 | 49.70
  Participants with >=50% Reductions | 42.80 | 34.50

10. Secondary Outcome: Percentage of Participants With Response to Treatment on Patient Global Impression-Improvement (PGI-I) at Endpoint
Description: PGI-I measures the participant's perception of improvement at the time of assessment compared with the start of treatment. Scores ranged from 1 (very much better) to 7 (very much worse). Response to treatment is defined by endpoint PGI rating of either "much better" or "very much better".The last observation carried forward (LOCF) method will be used for these analyses.
Time Frame: Week 13
Population: All participants who were randomized and had a baseline and at least 1 post-baseline observation.
Measure: Number; unit: percentage of participants
Arm/Group | 60 mg Duloxetine | Placebo
Number analyzed (Participants) | 194 | 196
percentage of participants
  Response to Treatment | 38.7 | 20.4
  1=Very much better | 3.10 | 2.60
  2=Much better | 35.60 | 17.90
  3=A little better | 40.70 | 51.00
  4=The same | 19.10 | 23.00
  5=A little worse | 1.50 | 3.60
  6=Much worse | 0.00 | 2.00
  7 = Very much worse | 0.00 | 0.00

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug. One participant in placebo arm did not receive study drug during the extension period.
Groups:
- 60 mg Duloxetine Double Blind: 60 mg duloxetine administered by mouth once a day (QD). Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD for 12 weeks.
- Placebo Double Blind: Placebo administered by mouth once a day (QD) for 13 weeks.
- 60 mg Duloxetine Extention: 60 mg duloxetine administered by mouth QD for 13 weeks.
- Placebo/60 mg Duloxetine Extention: 60 mg duloxetine administered by mouth QD for 13 weeks. Started on duloxetine 30 mg QD for 1 week and then titrated up to 60 mg duloxetine QD.
- 60 mg Duloxetine Taper: 1-week taper - participants taking 60 mg QD duloxetine during the study had their dosage reduced to 30 mg to minimize discontinuation-emergent adverse events (DEAEs).
- Placebo Taper: Taper Phase: 1-week taper - Placebo administered for 1 week if the participant discontinued from double blind treatment phase, or duloxetine 30 mg QD administered for 1 week if the participant discontinued from extension treatment phase or completed treatment. 1 week taper is to minimize discontinuation-emergent adverse events (DEAEs).
Arm/Group | 60 mg Duloxetine Double Blind | Placebo Double Blind | 60 mg Duloxetine Extention | Placebo/60 mg Duloxetine Extention | 60 mg Duloxetine Taper | Placebo Taper
Serious Adverse Events (participants affected / at risk) | 0/199 | 3/198 | 0/166 | 2/175 | 1/323 | 0/1
Other Adverse Events (participants affected / at risk) | 122/199 | 84/198 | 42/166 | 81/175 | 9/323 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 mg Duloxetine Double Blind (N=199) | Placebo Double Blind (N=198) | 60 mg Duloxetine Extention (N=166) | Placebo/60 mg Duloxetine Extention (N=175) | 60 mg Duloxetine Taper (N=323) | Placebo Taper (N=1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 60 mg Duloxetine Double Blind (N=199) | Placebo Double Blind (N=198) | 60 mg Duloxetine Extention (N=166) | Placebo/60 mg Duloxetine Extention (N=175) | 60 mg Duloxetine Taper (N=323) | Placebo Taper (N=1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 5 (7) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 21 (21) | 5 (5) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 31 (31) | 11 (11) | 3 (3) | 15 (15) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (25) | 5 (5) | 5 (5) | 8 (8) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Therapeutic response unexpected (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 7 (7) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 7 (8) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 3 (3) | 3 (3) | 10 (12) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 8 (9) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 16 (18) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/154 (0) | 0/148 (0) | 0/130 (0) | 1/129 (1) | 0/243 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 20 (21) | 9 (11) | 3 (3) | 7 (9) | 0 (0) | 0 (0)
Dreamy state (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 28 (31) | 10 (10) | 4 (4) | 10 (10) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 11 (11) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/45 (1) | 0/50 (0) | 0/36 (0) | 0/46 (0) | 0/80 (0) | 0/0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/45 (1) | 0/50 (0) | 0/36 (0) | 0/46 (0) | 0/80 (0) | 0/0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/154 (0) | 1/148 (1) | 0/130 (0) | 0/129 (0) | 0/243 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/154 (0) | 1/148 (1) | 0/130 (0) | 1/129 (1) | 0/243 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days